CLINICAL TRIAL: NCT00121498
Title: Preemptive Analgesia for Post Abdominal Hysterectomy Pain Management
Brief Title: Preemptive Analgesia for Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1571CTIL
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2004-12

CONDITIONS: Pain
Keywords: Pain; Hysterectomy; Preemptive; Lidocaine
MeSH Terms: conditions — Pain | interventions — Lidocaine; Anesthetics, Local

INTERVENTIONS:
Drug: Lidocaine (local anesthetics) 20 ml of 1 % subcutaneously

SUMMARY:
Preemptive analgesia is defined as "analgesic intervention provided before surgery to prevent or reduce subsequent pain". By preventing central sensitization using nociceptive blockers by regional analgesia we may able to produce a painless postsurgical state. The use of preemptive analgesia was reported in various surgical procedures, such as in limb surgeries, laparoscopic procedures, mastectomy and vaginal hysterectomy. Regarding abdominal hysterectomy there are only few reports, however both, malignancies and benign cases were included and conflicting results were obtained regarding the value of preemptive analgesia. Since hysterectomy is the most frequent major surgical procedure performed in gynecology, and it is estimated that by age 64 years, 40 % of women will have had a hysterectomy, it would be of great value to optimize pain treatment in these patients.

The aim of the present study was to evaluate the effectiveness of preemptive analgesia in women who undergo a transabdominal hysterectomy for benign uterine abnormalities.

Hypothesis: Lidocaine (5%) injection to the scar area before incision is effective in pain reduction among women who undergo a transabdominal hysterectomy for benign uterine abnormalities .

DETAILED DESCRIPTION:
Preemptive analgesia is defined as "analgesic intervention provided before surgery to prevent or reduce subsequent pain". By preventing central sensitization using nociceptive blockers by regional analgesia we may able to produce a painless postsurgical state. The use of preemptive analgesia was reported in various surgical procedures, such as in limb surgeries, laparoscopic procedures, mastectomy and vaginal hysterectomy. Regarding abdominal hysterectomy there are only few reports, however both, malignancies and benign cases were included and conflicting results were obtained regarding the value of preemptive analgesia. Since hysterectomy is the most frequent major surgical procedure performed in gynecology, and it is estimated that by age 64 years, 40 % of women will have had a hysterectomy, it would be of great value to optimize pain treatment in these patients.

The aim of the present study was to evaluate the effectiveness of preemptive analgesia in women who undergo a transabdominal hysterectomy for benign uterine abnormalities.

Material and Methods:

The study was approved by the Institutional Review Board in accordance with the Helsinki declaration. Rambam Medical Center is a public hospital, with no private patients and women are treated according to the same standard of guidelines. Women with a benign uterine myoma with or without menometrorrhagia are considered for the study. Patients are excluded if they have a systemic vascular or neurological disease, diabetes or more than two previous abdominal surgeries. A written informed consent, is obtained from the patients prior to randomization into two treatment groups. In the first group 20 ml of 1 % lidocaine were injected subcutaneously in the incisional region 15 minutes prior to the start of operation. In the second group 20 ml of normal saline are injected subcutaneously in the incisional area 15 minutes prior to operation. The syringes containing Lidocaine or Saline solution are prepared and coded by the pharmacist of the hospital. The surgeons, anesthetists and the nursing staff are all blinded to the type of solution, which is injected. The code is disclosed only at the end of the study. The anesthetic technique is standardized. A transverse lower abdominal incision is used in all patients. After completion of operation all patients are treated in the postoperative care unit for two hours. The time of arrival in the postoperative care unit is defined as time zero. Analgesia with morphine and pethidine was provided only on patient request. Thereafter patients are transferred to the Gynecological department.

The standard care for postoperative pain in our department is as follows: three fixed doses of Ibuprofen 400 mg at three hour intervals with the first dose administrated at arrival to the department (2 hours after operation). Women are informed, that they can receive a rescue dose of another medication for breakthrough pain if further analgesia is needed before the three hours elapses. In such cases they receive an intramuscular injection of 10 mg morphine. After completion of the fixed interval analgesic regimen, patients are allowed to receive four more doses of oral analgesics upon their request at 3-hour intervals. Starting from the second postoperative day, only oral analgesia is provided, on patient request. Pain intensity is evaluated in the first 24 postoperative hours, before the administration of each dose of analgesic medication. The self-report of pain is assessed by measurement on a 100 mm Visual Analogue Scale (VAS), ranging from "No Pain" (0), to "The most pain imaginable" (100). Patients are instructed to place a mark on the line that indicates the level of pain experienced. In addition, overall satisfaction with post surgical pain treatment was evaluated by patients 72 hours after surgery, with use of the same visual analogue scale but with phrasing of "very satisfactory" and "not satisfactory at all" The VAS results during the 24 hours and the number of doses of analgesia consumption during hospitalization will be compared between two groups using x test.

ELIGIBILITY:
Inclusion Criteria:

* Women who are scheduled for abdominal hysterectomy because of myomatous uterus via lower transverse incision.

Exclusion Criteria:

* Oncological disease
* Systemic vascular disease
* Neurological disease
* Diabetes
* More than two previous abdominal surgeries.

Ages: 35 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32
Dates: Start 2002-11; Study Completion 2003-09

PRIMARY OUTCOMES:
Postoperative pain scores: they were significantly lower in the study group in the first postoperative 8 hours

SECONDARY OUTCOMES:
No significant differences between the groups were noted in analgesic consumption on the second post- operative day

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jakobi, MD, Study Director — Department of OBGYN, Rambam Medical Center, Technion the Bruce Rappaort Faculty of Medicine
Locations (2):
- Israel (2):
  - Dept. OBGYN, Rambam Medical Center, Haifa
  - Rambam Medical Center, Dept OBGYN, Haifa

REFERENCES:
- [Result] Ali PB, Cotton BR, Williamson KM, Smith G. Intraperitoneal bupivacaine or lidocaine does not provide analgesia after total abdominal hysterectomy. Br J Anaesth. 1998 Feb;80(2):245-7. doi: 10.1093/bja/80.2.245. PMID 9602595